CLINICAL TRIAL: NCT00536185
Title: Variation in the ALOX5 Gene and Response to Omega-3 Fatty Acid Supplements
Brief Title: Heart & Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH); University of California, Davis (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); Alta Bates Summit Medical Center (Other); University of Southern California (Other)
Responsible Party: Charles Bolt Stephenson, PhD, Western Human Nutrition Resource Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R21AT003411-01A1 (NIH); R21AT003411-01A1 (NIH)
Record Dates: First submitted 2007-09-05; First posted 2007-09-27 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Heart Disease
Keywords: ALOX5; 5-lipoxygenase; Heart Disease; Blacks
MeSH Terms: conditions — Heart Diseases | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Fish Oil
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — capsules, 5.0 g/d fish oil concentrate (3.0 g/d EPA + DHA), 6 weeks
  Arms: 1
Dietary Supplement: Placebo — capsule, 5.0 g/d corn/soybean oil (50/50 mixture), 6 weeks
  Arms: 2

SUMMARY:
We hope to learn more about why certain people have higher levels of the 5-LO protein and whether taking fish oil supplements gives such individuals greater protection than others against cardiovascular disease. The 5-LO protein is important in the development of heart disease because it converts a type of oil from meat into a compound that can cause inflammation in blood vessels. This inflammation is a major cause of heart disease.

Researchers think that people with higher levels of a protein called 5-LO in their white blood cells may have a healthier response to using fish oil supplements than do people with lower levels of this protein.

DETAILED DESCRIPTION:
Fish oil supplements will be given to subjects with different variants in the promoter region of the arachidonate 5-lipoxygenase (ALOX5) gene and outcome measures will be evaluated after 6 wk of supplementation. These outcomes include ALOX5 protein levels (also called 5-lipoxygenase, or 5-LO), leukotriene levels, markers of inflammation, and blood lipids. The 5-LO enzyme converts arachidonic acid (AA) to leukotrienes that promote inflammation. Subjects with different promoter variants are hypothesized to have different basal or stimulated levels of 5-LO expression. Preliminary data suggests that subjects with a promoter variant that causes increased 5-LO expression also may have a "better" anti-inflammatory or lipid-lowering response to fish oil supplements. The homozygous variant genotype is much more common in African Americans than other groups thus we propose to conduct the study in African Americans. The fish oil eicosapentaenoic acid (EPA) competitively inhibits conversion of AA to pro-inflammatory 4-series leukotrienes.

The grant proposes to conduct a community-based, double-masked, randomized, placebo-controlled trial; n = 15/group, total = 166 (genotypes 44 will have n = 8). The intervention group will receive 5.0 g/d fish oil concentrate (3.0 g/d EPA + DHA) for 6 wk. The study will be conducted in Oakland, Davis, and Sacramento, California where African Americans 20 - 59 y of age without serious chronic disease will be recruited.

A recent observational study indicates that subjects with a variant allele for ALOX5 may be at greater risk for cardiovascular disease and, at the same time, may derive a greater benefit from omega-3 fatty acid supplements than do subjects homozygous for the common allele. The variant alleles are less common in the white population (18%) than in the black population (52%). Since African Americans have a higher prevalence of cardiovascular disease and of the ALOX5 variant alleles, as shown in epidemiologic studies, they may have a greater benefit from omega-3 supplementation in the reduction of inflammation and cardiovascular risk factors. Recruitment will be conducted through the community service, Ethnic Health Institute (EHI), of Alta Bates Summit Medical Center in conjunction with UCD, and outreach efforts from the USDA, ARS, Western Human Nutrition Research Center (WHNRC) at UC Davis. We will determine if subjects with one or two variant ALOX5 alleles have higher ALOX5 gene expression, higher production of AA-derived leukotrienes, and a better response to omega-3 supplements than do subjects homozygous for the common allele.

ELIGIBILITY:
Inclusion Criteria:

* African-American, Black, or persons of African Descent
* Generally Healthy
* 20 - 59 years of age

Exclusion Criteria:

* Chronic Diseases (Heart disease, cancer, diabetes, etc.)
* Smoke > 14 cigarettes per week
* Consume > 14 alcoholic drinks per week
* Pregnant Women

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
(a) ALOX5 mRNA and protein in resting and stimulated cultures of purified monocytes and purified granulocytes (b) Arachidonic acid-derived leukotrienes in resting and stimulated cultures of whole blood, purified monocytes and purified granulocytes | 6 weeks

SECONDARY OUTCOMES:
Proinflammatory cytokines, C-reactive protein, triglycerides, glucose and insulin in plasma, and resting heart rate and blood pressure | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Stephensen, PhD, Principal Investigator — UC Davis & U.S. Department of Agriculture
Locations (3):
- United States (3):
  - UC Davis, Western Human Nutrition Research Center, Davis, California
  - Ethnich Health Institute, Oakland, California
  - UC Davis (TICON-1), Sacramento, California

REFERENCES:
- [Derived] O'Sullivan A, Armstrong P, Schuster GU, Pedersen TL, Allayee H, Stephensen CB, Newman JW. Habitual diets rich in dark-green vegetables are associated with an increased response to omega-3 fatty acid supplementation in Americans of African ancestry. J Nutr. 2014 Feb;144(2):123-31. doi: 10.3945/jn.113.181875. Epub 2013 Nov 20. PMID 24259553
- [Derived] Armstrong P, Kelley DS, Newman JW, Staggers FE Sr, Hartiala J, Allayee H, Stephensen CB. Arachidonate 5-lipoxygenase gene variants affect response to fish oil supplementation by healthy African Americans. J Nutr. 2012 Aug;142(8):1417-28. doi: 10.3945/jn.112.159814. Epub 2012 Jun 27. PMID 22739369
- [Derived] Vikman S, Brena RM, Armstrong P, Hartiala J, Stephensen CB, Allayee H. Functional analysis of 5-lipoxygenase promoter repeat variants. Hum Mol Genet. 2009 Dec 1;18(23):4521-9. doi: 10.1093/hmg/ddp414. Epub 2009 Aug 28. PMID 19717473
- See also: Western Human Nutrition Research website — http://www.ars.usda.gov/main/site_main.htm?modecode=53062500